CLINICAL TRIAL: NCT00725842
Title: Relapse Rate and Predictive Factors in the Treatment of Hepatitis C in Common Clinical Practice
Brief Title: Relapse Rate in Hepatitis C Patients Treated With Peginterferon Alfa-2b Plus Ribavirin in Common Clinical Practice in France (P05484)(Completed)
Acronym: RE-CHUT
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05484
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C; Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peg-IFN alfa-2b + ribavirin: Participants with chronic hepatitis C (CHC) treated with Peg-IFN alfa-2b + ribavirin as first treatment, in common clinical practice, who had negative hepatitis-C virus (HCV)-ribonucleic acid (RNA) by the end of treatment (24 or 48 weeks per product labeling).
  Interventions: Biological: Peg-IFN alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Biological: Peg-IFN alfa-2b — Peg-IFN alfa-2b administered in accordance with approved labeling
  Other Names: SCH 054031
Drug: Ribavirin — Ribavirin administered in accordance with approved labeling
  Other Names: SCH 018908

SUMMARY:
The objective of this study is to determine the relapse rate in the French patient population with chronic hepatitis C (CHC) previously treated with PegInterferon Alfa-2b (Peg-IFN alfa-2b) plus Ribavirin according to standard clinical practice. Treatment was to be completed prior to the enrollment in the current study. The study will also aim to identify factors that are predictive of relapse. Relapse rate is defined as the percentage of patients with negative viral load at end of treatment who again have positive viral load at 6 months after the end of treatment.

DETAILED DESCRIPTION:
Non-probability sampling: The study population consists of adult patients over the age of 18 affected by CHC who were previously treated for the first time with Peg-IFN alfa-2b plus ribavirin and achieved end-of-treatment response. Five hundred ninety patients must be recruited in order to evaluate the objectives of the study. The patients must meet all inclusion criteria and not meet any of the exclusion criteria in order to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* The patient must demonstrate his/her continued willingness to participate in the study.
* The patient must be at least 18 years of age, of either gender.
* Patients with chronic hepatitis C (any genotype) who received Peg-IFN alfa-2b + Ribavirin as first treatment for hepatitis C.
* Negative HCV-RNA at the end of treatment (24 or 48 weeks according to the product labeling as appropriate), measured by the assay used at each institution. Only institutions using an assay with a limit of detection of 50 IU/mL or less will be eligible.

Exclusion Criteria:

* Patients who completed treatment with PegInterferon Alfa-2b plus Ribavirin more than 4 weeks before study entry.
* Patients with positive HCV-RNA at the end of treatment (24 or 48 weeks according to the product labeling as appropriate).
* Patients treated for a period shorter than the enrollment period.
* Patients co-infected with human immunodeficiency virus (HIV).
* Patients co-infected with hepatitis B virus (HBV).
* Patients who do not use appropriate effective method of birth control after the end of treatment (according to legal recommendations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatitis C previously treated with Peg-IFN alfa-2b + ribavirin in common clinical practice at approximately 60 centers in France.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peg-IFN Alfa-2b + Ribavirin
Started | 97
Participants Eligible for Analysis | 90
Completed | 57
Not Completed | 40
Not completed — Lost to Follow-up | 19
Not completed — Death | 1
Not completed — Positive HCV-RNA at Visit 2 | 13
Not completed — Consent date prior to study start date | 5
Not completed — Inclusion criterion not met | 1
Not completed — No Visit 1 data | 1

BASELINE CHARACTERISTICS:
Arm/Group | Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] — Age data unavailable for the 7 participants excluded from analysis.
  years | 46.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender data unavailable for the 7 participants excluded from analysis.
  Participants
    Female | 25
    Male | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Hepatitis C Virus (HCV)-Ribonucleic Acid (RNA) at 24 Weeks Off-treatment
Description: HCV-RNA virus levels were measured by polymerase chain reaction (PCR) assay 24 weeks post end of treatment (EOT) with Peg-IFN alfa-2b + ribavirin. Participants with positive HCV-RNA were considered relapsers.
Time Frame: 24 weeks post end of treatment (EOT)
Population: Of the 97 participants who started the study, 7 were excluded from analysis because of protocol violations. 90 participants underwent HCV-RNA testing at Week 24 post EOT.
Measure: Number; unit: participants
Arm/Group | Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 90
participants | 13

2. Secondary Outcome: Number of Participants With Rapid Virologic Response (RVR), Early Virologic Response (EVR), or Slow Response Who Relapsed After Treatment
Description: Negative HCV-RNA at Week 4 of treatment with Peg-IFN alfa-2b + ribavirin was considered RVR; negative HCV-RNA at Week 12 of treatment with Peg-IFN alfa-2b + ribavirin was considered EVR; negative HCV-RNA between Week 12 and the end of treatment with Peg-IFN alfa-2b + ribavirin was considered a slow response. For participants who achieved RVR, EVR, or slow response, the relapse rate at 24 Weeks post EOT was to be determined on this observational study; relapse was defined as positive HCV-RNA.
Time Frame: 24 weeks post EOT
Population: The planned analysis for this outcome measure was not performed due to insufficient enrollment.
Arm/Group | Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 0

3. Secondary Outcome: Assessment of Pre-treatment Risk Factors of Relapse in Participants With Sustained Virologic Response
Description: Baseline risk factors included but were not limited to viral load, genotype 1a versus 1b, histology, treatment compliance, gender, age, and substance abuse. Sustained virologic response was defined as having negative HCV-RNA at 24 weeks post EOT. Relapse was defined as positive HCV-RNA.
Time Frame: Baseline and 24 weeks post EOT
Population: The planned analysis for this outcome measure was not performed due to insufficient enrollment.
Arm/Group | Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Positive HCV-RNA at 72 Weeks Off-treatment
Description: HCV-RNA virus levels were measured by polymerase chain reaction (PCR) assay 72 weeks post EOT with Peg-IFN alfa-2b + ribavirin. Participants with positive HCV-RNA at Week 72 post EOT were considered late relapsers.
Time Frame: 72 weeks post EOT
Population: 77 of 90 participants had a negative HCV-RNA at Week 24 post EOT. These 77 were then evaluated for relapse at Week 72 post EOT.
Measure: Number; unit: participants
Arm/Group | Peg-IFN Alfa-2b + Ribavirin
Number analyzed (Participants) | 77
participants | 3

ADVERSE EVENTS:
Description: The safety data set included 96 of the 97 participants who started on study; no safety data were available for 1 participant.
Arm/Group | Peg-IFN Alfa-2b + Ribavirin
Serious Adverse Events (participants affected / at risk) | 5/96
Other Adverse Events (participants affected / at risk) | 21/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peg-IFN Alfa-2b + Ribavirin (N=96)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Death (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peg-IFN Alfa-2b + Ribavirin (N=96)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Asthenia (General disorders) | 15 (16)

LIMITATIONS AND CAVEATS:
Due to low enrollment some planned analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study data disclosure is prohibited; data and study results are the exclusive property of the Sponsor.